CLINICAL TRIAL: NCT05512702
Title: Treatment Approach in Patients Diagnosed With Pulmonary Thromboembolism With Intermediate-High Risk Interms of Early Mortality After the Establisment of Ege Pulmonary Embolism Team
Brief Title: Reduced Dose Thrombolytic in Intermediate/High Risk Pulmonary Thromboembolism
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Pervin KORKMAZ, Associated Professor, Ege University
Other Study IDs: 21-AKD-107
Record Dates: First submitted 2022-08-22; First posted 2022-08-23 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Pulmonary Embolism
Keywords: Pulmonary Embolism; Pulmonary Embolism Response Teams; Thrombolytic Treatment; Anticoagulation Treatment; Mortality; Complication
MeSH Terms: conditions — Pulmonary Embolism | interventions — Tissue Plasminogen Activator; Dalteparin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Thrombolytic Treatment Group: These are the patients with intermediate-high riskPE and consulted by EGEPET. They received reduced dose thrombolytic treatment.
  Interventions: Drug: Tissue Plasminogen Activator, Alteplase
- Anticoagulation Treatment Group: This group includes patients who diagnosed wit PE before the establishment of EGEPET. And these patients are classed into intermediate-high risk based on early mortality and received anticoagulation treatment, not thrombolytic treatment.
  Interventions: Drug: Low-molecular weight heparin

INTERVENTIONS:
Drug: Tissue Plasminogen Activator, Alteplase — Reduced dose (50 mg) Alteplase is used for the patients in the thrombolytic treatment group.
  Groups: Thrombolytic Treatment Group
Drug: Low-molecular weight heparin — Patients in the anticoagulation treatment group receive this treatment and do not receive thrombolytic treatment.
  Groups: Anticoagulation Treatment Group

SUMMARY:
Pulmonary Embolism(PE) requires multidisciplinary approach as a highly morbid and mortal disease. This multidisciplinary approach creates clinical benefits in diagnostic and therapeutic process. And these benefits are pointed out in certain studies and guidelines. For these reasons, a Pulmonary Embolism Response Team (PERT) was established on 5 th November 2018 which is called as Ege Pulmonary Embolism Team (EGEPET) in our university.

In recent years, it is stated that the carefully use of thrombolytic in patients with intermediate-high risk PE based on early mortality classification. Some studies have reported that the use of thrombolytic may cause clinical benefits. But which used drug and which dose are not defined clearly yet.

After establishment of EGEPET, the investigators observed that patients with intermediate-high risk PE more receive reduced dose thrombolytic than the pre-EGEPET period. And the investigators aimed to compare treatment changes after and before the establishment of EGEPET. Also, the investigator will compare initial reduced dose thrombolytic therapy after EGEPET with initial anticoagulation therapy before EGEPET (historical group) in terms of mortality and complication.

As the reduced dose thrombolytic, Alteplase 50 mg is used in our hospital. Low-molecular weight heparin (LMWH), standard heparin and rarely Fondaparinux are used for anticoagulation therapy. Low-molecular weight heparin is generally applied for treatment, in case there is no contraindication.

Our primary end-point is to assess 30-day mortality and secondary-end points are to detect in one year-mortality and complications. The investigators will compare the mortality and complication rates in these groups.

N0 hypothesis; In the intermediate-high risk group diagnosed with PE, there is an increased mortality rate in the patients treated with half-dose thrombolytic (Alteplase 50 mg) than our historical group or the literature.

N1 hypothesis; In the intermediate-high risk group diagnosed with PE, there is no an increased mortality rate in the patients treated with half-dose thrombolytic (Alteplase 50 mg) than our historical group or the literature.

DETAILED DESCRIPTION:
Pulmonary thromboembolism ranks 3rd among cardiovascular diseases in terms of mortality. Pulmonary Embolism (PE) is a challenging disease that requires rapid approach both in the diagnosis and treatment process. Due to the challenging nature of the disease, Pulmonary Embolism Response Teams (PERT) have emerged for quick intervention in patients with PE. In the management of PE, multidisciplinary approach that includes the branches of pulmonary diseases, cardiology, emergency medicine, cardiovascular surgery, anesthesiology and radiology provides clinical advantages. Therefore, a PERT was established and called Ege Pulmonary Embolism Team (EGEPET). EGEPET established on 5th of November 2018. This team contains specialists from Pulmonary Diseases, Cardiology, Emergency Medicine, Cardiovascular Surgery, Anesthesiology and Radiology Departments. EGEPET works during 7/24 as a response team. It has been stated in recent publications and pulmonary thromboembolism guidelines that the establishment of multidisciplinary study group which is similar to our group will be more effective in the diagnosis, treatment and follow-up processes of PE patients.

Specially, there are some different opinions for the treatment of Intermediate-High risk based on according to early mortality with PE patients. While some guidelines suggest initial anticoagulation treatment without thrombolytic treatment, some researchers state that thrombolytic treatment can be used in Intermediate-High risk patients. These researchers indicate that the careful use of thrombolytic can be improved in clinical situation of PE patients. The careful usage is meant to use reduced dose thrombolytic and to follow up the patients closely for bleeding complication.

In cases diagnosed with intermediate-high risk PE in related to early mortality, it has been seen that half-dose thrombolytics are given mostly in our daily life practice after EGEPET.

So, the investigators planned to evaluate the mortality and morbidity rates in the patients who were diagnosed with pulmonary thromboembolism with intermediate-high risk in terms of early mortality and who received half-dose thrombolytics according to the result of the EGEPET consultation.

50 mg Alteplase is used as thrombolytic treatment and, low-molecular weight heparin (LMWH), standard heparin and rarely Fondaparinux are used for initial anticoagulation treatment. Low-molecular weight heparin is generally applied for treatment, in case there is no contraindication.

This study is an observational drug study. Researchers of this study did not and will not intervene the treatment of patients. Treatment decision of the patients is decided by EGEPET physicians.

The investigators will compare the patients diagnosed with intermediate-high risk PE who received reduced dose thrombolytic which the decision is made by EGEPET with the other patients who did not get thrombolytic treatment in terms of mortality and morbidity.

The other patient group with intermediate-high risk PE will be created from our historical data to prevent to selection bias. Because, EGEPET offers generally reduced dose thrombolytic in intermediate-high risk PE patients. Otherwise, patients having high bleeding scores (e.g. RIETE bleeding score), multiple and severe comorbidities or patients who are quite old generally receive only anticoagulation treatment.

The patients assessed our study were classed into three groups. All of the patients have PE and are stated into intermediate-high risk according to early mortality.

First group is prospective group, which contains patients recruited after approval of ethic committee of this study. Ethic committee was taken from both organization Ege University and The Ministry of Health-Türkiye.

Second group is retrospective group, which contains patients evaluated by EGEPET and received reduced dose thrombolytic treatment.

Third group is called as historical control group. This patients group were diagnosed and treated with anticoagulants not thrombolytic treatment before establishment of EGEPET.

First and second groups compose the thrombolytic group, third group create the anticoagulant group (control)

The investigators are going to collect data (clinical, laboratory and radiological variables) of these patients to get detailed clinical information.

The investigators will compare the thrombolytic group with anticoagulant group (control). The primary end-point is to evaluate 30-day mortality and secondary-end point are to detect in one year-mortality and complications.

The investigators will compare mortality and complication rates in both groups.

N0 hypothesis; In the intermediate-high risk group diagnosed with PE, there is an increased mortality rate in the patients treated with half-dose thrombolytic (Alteplase 50 mg) than our historical group or the literature.

N1 hypothesis; In the intermediate-high risk group diagnosed with PE, there is no an increased mortality rate in the patients treated with half-dose thrombolytic (Alteplase 50 mg) than our historical group or the literature.

ELIGIBILITY:
Inclusion Criteria:

* Patients which are in intermediate-high risk class ased on mortality in the ESC/ERS Pulmonary Embolism Risk Classification

Exclusion Criteria:

* Unwillingness of patient to participate in the study
* The case is in the intermediate-high risk class, but there is an unstable disease that will affect mortality due to malignancy or general medical condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this study, intermediate-high risk PE patients will divide whether receice thrombolytic treatment or not. And two group are going to compare in the context of mortality rate. We anticipate that 50 patients should be enough for statistically powerful study. We predict this number according to previous studies and power analyses.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-06-03 (Actual); Primary Completion 2023-06-03 (Estimated); Study Completion 2024-06-03 (Estimated)

PRIMARY OUTCOMES:
30 day Mortality | 30 day after diagnosis of pulmonary tromboembolism
  Includes 30-day mortality and contains all causes of death.

SECONDARY OUTCOMES:
1 year Mortality | 1 year after diagnosis of pulmonary tromboembolism
  Includes 1 year mortality and contains all causes of death.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University, Izmir, Bornova/İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mirambeaux R, Leon F, Bikdeli B, Morillo R, Barrios D, Mercedes E, Moores L, Tapson V, Yusen RD, Jimenez D. Intermediate-High Risk Pulmonary Embolism. TH Open. 2019 Dec 4;3(4):e356-e363. doi: 10.1055/s-0039-3401003. eCollection 2019 Oct. PMID 31815247
- [Background] Konstantinides SV, Meyer G, Becattini C, Bueno H, Geersing GJ, Harjola VP, Huisman MV, Humbert M, Jennings CS, Jimenez D, Kucher N, Lang IM, Lankeit M, Lorusso R, Mazzolai L, Meneveau N, Ni Ainle F, Prandoni P, Pruszczyk P, Righini M, Torbicki A, Van Belle E, Zamorano JL; ESC Scientific Document Group. 2019 ESC Guidelines for the diagnosis and management of acute pulmonary embolism developed in collaboration with the European Respiratory Society (ERS). Eur Heart J. 2020 Jan 21;41(4):543-603. doi: 10.1093/eurheartj/ehz405. No abstract available. PMID 31504429
- [Background] Sharifi M, Bay C, Skrocki L, Rahimi F, Mehdipour M; "MOPETT" Investigators. Moderate pulmonary embolism treated with thrombolysis (from the "MOPETT" Trial). Am J Cardiol. 2013 Jan 15;111(2):273-7. doi: 10.1016/j.amjcard.2012.09.027. Epub 2012 Oct 24. PMID 23102885
- [Background] Meyer G, Vicaut E, Danays T, Agnelli G, Becattini C, Beyer-Westendorf J, Bluhmki E, Bouvaist H, Brenner B, Couturaud F, Dellas C, Empen K, Franca A, Galie N, Geibel A, Goldhaber SZ, Jimenez D, Kozak M, Kupatt C, Kucher N, Lang IM, Lankeit M, Meneveau N, Pacouret G, Palazzini M, Petris A, Pruszczyk P, Rugolotto M, Salvi A, Schellong S, Sebbane M, Sobkowicz B, Stefanovic BS, Thiele H, Torbicki A, Verschuren F, Konstantinides SV; PEITHO Investigators. Fibrinolysis for patients with intermediate-risk pulmonary embolism. N Engl J Med. 2014 Apr 10;370(15):1402-11. doi: 10.1056/NEJMoa1302097. PMID 24716681
- [Result] Wendelboe AM, Raskob GE. Global Burden of Thrombosis: Epidemiologic Aspects. Circ Res. 2016 Apr 29;118(9):1340-7. doi: 10.1161/CIRCRESAHA.115.306841. PMID 27126645